CLINICAL TRIAL: NCT01917019
Title: A Multicenter, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Safety and Efficacy of Oral Prolonged-Release Fampridine (BIIB041) in Japanese Subjects With Multiple Sclerosis Followed by an Open-Label Safety Extension
Brief Title: A Safety and Efficacy Study of Oral Prolonged-Release Fampridine (BIIB041) in Japanese Participants With Multiple Sclerosis
Acronym: MOTION - JAPAN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 218MS304
Record Dates: First submitted 2013-08-02; First posted 2013-08-06 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Multiple Sclerosis, Remittent Progressive; Multiple Sclerosis, Primary Progressive; Relapsing-Remitting Multiple Sclerosis; Secondary Progressive Multiple Sclerosis; Multiple Sclerosis
Keywords: Japan
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — 4-Aminopyridine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- Part A Placebo (Placebo Comparator): Part A: All participants will receive placebo orally twice daily for the first 2 weeks and then be randomized to receive prolonged-release fampridine 10 mg or matching placebo tablets orally twice daily for up to 14 weeks.
  Interventions: Drug: Placebo
- Part A prolonged-release fampridine (Experimental): Part A: All participants will receive placebo orally twice daily for the first 2 weeks and then be randomized to receive prolonged-release fampridine 10 mg or matching placebo tablets orally twice daily for up to 14 weeks.
  Interventions: Drug: BIIB041 (fampridine)
- Part B prolonged-release fampridine (Experimental): Part B: Eligible participants will receive open label treatment with prolonged-release fampridine 10mg orally twice daily for up to 52 weeks.
  Interventions: Drug: BIIB041 (fampridine)
- Part C prolonged-release fampridine (Experimental): Part C: Eligible participants will receive open label treatment with prolonged-release fampridine 10mg orally twice daily until marketed product is available.
  Interventions: Drug: BIIB041 (fampridine)

INTERVENTIONS:
Drug: Placebo — matching placebo tablets
  Arms: Part A Placebo
Drug: BIIB041 (fampridine) — fampridine prolonged-release tablets
  Other Names: Fampyra; prolonged-release fampridine; dalfampridine; Ampyra
  Arms: Part A prolonged-release fampridine; Part B prolonged-release fampridine; Part C prolonged-release fampridine

SUMMARY:
This is a multicenter study conducted in 3 parts. Part A is a double-blind placebo-controlled parallel-group period, and Part B and C are open-label extension periods. The primary objective of the double-blind study (Part A) is to assess the effect of Prolonged-Release Fampridine treatment on walking speed as measured by the T25FW (timed 25 foot walk) in Japanese participants with Multiple Sclerosis. The secondary objective of the double-blind portion of the study is to evaluate the safety and tolerability of prolonged-release Fampridine in this study population. The primary objective of the open-label extension study (Part B) is to evaluate the long-term safety profile of prolonged-release Fampridine. The primary objective of the additional open-label extension (Part C) is to provide participants who complete the study with continued access to prolonged-release fampridine until marketed drug can be used at the applicable site or until sponsor decision to discontinue the study.

ELIGIBILITY:
Key Inclusion Criteria:

Part A

To be eligible to participate in Part A, candidates must meet the following eligibility criteria at screening or at the timepoint specified in the individual eligibility criterion listed (potential subjects who fail screening may be rescreened 1 time):

1. Must have a diagnosis of primary-progressive, secondary progressive, progressive relapsing, or relapsing-remitting MS as defined by the revised McDonald Committee criteria ([Lublin and Reingold 1996; McDonald 2001; Polman 2005]) of at least 2 months duration.
2. Must be able to complete the T25FW with or without a walking aid in 8 to 45 seconds at the screening visit.

Part B

To be eligible to participate in Part B, candidates must meet the following criteria at the Week 21 visit in Part A, which is the first visit for Part B:

1. Completed all visits in Part A of the study.

Part C

To be eligible to participate in Part C, candidates must meet the following criteria at the Week 52 visit in Part B, which is the first visit for Part C:

1. Completed all visits in Part B of the study.

Key Exclusion Criteria:

1. Known allergy to pyridine-containing substances, or any of the inactive ingredients of the prolonged-release fampridine tablet
2. Any prior history of seizures, epilepsy, or other convulsive disorder, with the exception of febrile seizures in childhood, or prior history of epileptiform activity on electroencephalogram.
3. Any form of renal impairment as defined by a creatinine clearance (CrCl) of <80 mL/min (estimated by the central laboratory).
4. Known history of cardiac arrhythmia or cardiac conduction disorders requiring medical or surgical intervention, or any clinically significant ECG abnormality (as determined by the Investigator) at the screening visit or Day 1.
5. Any prior treatment with fampridine (4 AP) or 3,4 diaminopyridine in any formulation.
6. Treatment with an investigational drug or approved therapy for investigational use within 30 days (or 5 half lives, whichever is longer) prior to the screening visit.
7. Participation in an investigational study (with the exception of observational studies) within 30 days prior to the screening visit or plans to enroll in another interventional investigational study at any time during this study.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2013-08; Primary Completion 2015-10 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
The proportion of participants who show a consistent improvement in walking speed | Part A (Up to 21 Weeks)
Number of participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Part B (54 Weeks)

SECONDARY OUTCOMES:
Number of participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Part A (Up to 21 Weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (19):
- Japan (19):
  - Research Site, Bunkyō City
  - Research Site, Chiba
  - Research Site, Fuchū
  - Research Site, Fukuoka
  - Research Site, Kawagoe-shi
  - Research Site, Kodaira-shi
  - Research Site, Kyoto
  - Research Site, Morioka
  - Research Site, Niigata
  - Research Site, Obihiro
  - Research Site, Osaka
  - Research Site, Ōta-ku
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Shinjuku-ku
  - Research Site, Suita-shi
  - Research Site, Toon-shi
  - Research Site, Ube-shi
  - Research Site, Yachiyo-shi